CLINICAL TRIAL: NCT04470245
Title: Cubital Tunnel Syndrome and Diffusion Tensor Magnetic Resonance Imaging: A Proof of Concept Study
Brief Title: Cubital Tunnel Syndrome and Diffusion MRI: A Proof of Concept Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PL19/122843
Record Dates: First submitted 2020-07-08; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Cubital Tunnel Syndrome
MeSH Terms: conditions — Cubital Tunnel Syndrome | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Active Comparator)
  Interventions: Diagnostic Test: magnetic resonance imaging (MRI)
- Patients undergoing surgery (Active Comparator): We will include adults (over 18 years of age) undergoing surgical decompression of the ulnar nerve at the elbow for cubital tunnel syndrome.
  Interventions: Diagnostic Test: magnetic resonance imaging (MRI)

INTERVENTIONS:
Diagnostic Test: magnetic resonance imaging (MRI) — Our study will include healthy volunteers (to refine the scanning sequence) and patients undergoing surgery for CTS. Patients will be scanned before and after their operation using cutting-edge diffusion MRI techniques.

SUMMARY:
Cubital Tunnel Syndrome (CTS) results from compression of the ulnar nerve at the elbow (colloquially termed the "funny bone"). CTS affects up to 6% of the population and 6000 patients undergo surgery annually in the UK. Surgery is the only proven treatment for CTS, although up to 30% of patients do not improve. Therefore, there is a pressing need to develop a reliable test to diagnose CTS to improve the selection of patients for surgery.

New techniques in the field of magnetic resonance imaging (MRI) allow the visualisation of nerve structure and function. Diffusion tensor MRI, also known as diffusion tensor imaging (DTI), can diagnose CTS with superior diagnostic accuracy and could enable the reliable diagnostic of CTS, improving the selection of patients for surgery.

The study will include healthy volunteers (to refine the scanning sequence) and patients undergoing surgery for CTS. Patients will be scanned preoperatively and postoperatively using cutting-edge diffusion MRI techniques. The primary outcome will be change in the MRI-derived diffusion metrics following surgery. Secondary outcomes will consider how MRI relates to patient-reported outcomes and conventional clinical tests (ultrasound and nerve conduction studies).

Leeds is the ideal location for this research because a) Leeds institutions are the most highly cited organisations in musculoskeletal research, b) Leeds houses the National Centre for Hyperpolarized MRI and a state-of-the-art MRI scanner, and c) Leeds is an internationally recognised centre of excellence for complex upper limb surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 years of age) undergoing surgical decompression of the ulnar nerve at the elbow for cubital tunnel syndrome.

Exclusion Criteria:

* Unable to get into the MRI scanner due to habitus or claustrophobia
* Unable to lie still due to any cause (eg. athetoid movements, dystonias, chorea, etc)
* Intraocular or intracranial metallic foreign bodies
* Active implants (eg. pacemakers, implantable cardiac defibrillators, nerve stimulators, etc) which are not MRI safe or conditional.
* Pregnancy - whilst there are no known adverse effects of MRI16-18 to the mother or fetus, MRI is generally avoided in pregnancy due to the acoustic trauma19 and inductive heating generated by alternating magnetic fields.
* Any metallic implants in the elbow

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
The question is whether the MRI diffusion metrics of the ulnar nerve in patients with the cubital tunnel | 60 minutes
  change following surgical decompression.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom